CLINICAL TRIAL: NCT01969422
Title: Online Question-answering and Conventional Consultation With a Dermatologist
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-0340
Record Dates: First submitted 2013-10-10; First posted 2013-10-25 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Skin Diseases
MeSH Terms: conditions — Skin Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- observation group: observation
  Interventions: Procedure: observation

INTERVENTIONS:
Procedure: observation — intervention is the contact with online question answering serice ad subseudd

SUMMARY:
Comparison of online question-answering system and conventional consultation for dermatological questions:

* same diagnosis?
* same information, which had been collected?
* same recommendations about treatment?
* what were the relevant differences of the two?

DETAILED DESCRIPTION:
mainly, ICD codes and dermatological diagnosis codes according to the AAD will be used.

ELIGIBILITY:
Inclusion criteria:

- a conventional dermatological consultation after a question in the online question-answering system.

Exclusion criteria:

-power of veto after information of patient

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: persons with a question on skin disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Correlation of online and clinical diagnosis by Spearman's Rho | physical consultation date

CONTACTS AND LOCATIONS:
Overall Officials: Guenther Hofbauer, Prof MD, Principal Investigator — University Hospital Zurich, Department of Dermatology
Locations (1):
- University Hospital Zurich, Department of Dermatology, Zurich, Canton of Zurich, Switzerland